CLINICAL TRIAL: NCT06166368
Title: the Bispebjerg Study of Diurnal Variations
Acronym: DIURNAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Henriette P. Sennels, MD PhD., Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Diurnal variations
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Diurnal
MeSH Terms: interventions — Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diurnal variations (Experimental): Venous blood samples were obtained under standardized conditions from 24 healthy young men every third hour through 24 hours
  Interventions: Other: Diurnal variation

INTERVENTIONS:
Other: Diurnal variation — Venous blood samples were obtained under standardized circumstances from 24 healthy young men every third hour through 24 hours, nine time points in total.

SUMMARY:
To evaluate the influence of time of day on the circulating concentrations of various biochemical markers in healthy men

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Normal sleep-wake pattern

Exclusion Criteria:

* acute or chronic medical diseases
* had worked nightshifts the last 14 days before the study
* transatlantic traveling the last 14 days before the study
* had been smoking the last 14 days before the study
* had an irregular sleep-wake pattern,
* didn't sleep 7-8 hours pr night
* were extreme morning- or evening types,
* had plasma hemoglobin < 8.0 mmol/L
* ody mass index (BMI) <18.5 kg/m2 or >24.9 kg/m2.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10-11 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-01-01 (Actual)

PRIMARY OUTCOMES:
hematology parameters | 24 hours
  Composite measurement of hematological measurements

SECONDARY OUTCOMES:
Plasma Levels of Glucagon | 24 hours
Plasma levels of GLP-1 | 24 hours
Plasma levels of GIP | 24 hours
Plasma levels of c-peptide | 24 hours
Plasma levels of glucose | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Henriette P Sennels, MD PhD, Principal Investigator — Bispebjerg Hospital

IPD SHARING:
Plan to Share IPD: No
Not allowed by ethical committe

REFERENCES:
- [Background] Sennels HP, Jorgensen HL, Hansen AL, Goetze JP, Fahrenkrug J. Diurnal variation of hematology parameters in healthy young males: the Bispebjerg study of diurnal variations. Scand J Clin Lab Invest. 2011 Nov;71(7):532-41. doi: 10.3109/00365513.2011.602422. PMID 21988588
- [Background] Goetze JP, Jorgensen HL, Sennels HP, Fahrenkrug J. Diurnal plasma concentrations of natriuretic propeptides in healthy young males. Clin Chem. 2012 Apr;58(4):789-92. doi: 10.1373/clinchem.2011.178921. Epub 2012 Jan 26. No abstract available. PMID 22282468
- [Background] Sennels HP, Jorgensen HL, Goetze JP, Fahrenkrug J. Rhythmic 24-hour variations of frequently used clinical biochemical parameters in healthy young males--the Bispebjerg study of diurnal variations. Scand J Clin Lab Invest. 2012 Jul;72(4):287-95. doi: 10.3109/00365513.2012.662281. Epub 2012 Mar 8. PMID 22397709
- [Background] Timm A, Fahrenkrug J, Jorgensen HL, Sennels HP, Goetze JP. Diurnal variation of von Willebrand factor in plasma: the Bispebjerg study of diurnal variations. Eur J Haematol. 2014 Jul;93(1):48-53. doi: 10.1111/ejh.12298. Epub 2014 Mar 18. PMID 24571735
- [Background] Sennels HP, Jorgensen HL, Fahrenkrug J. Diurnal changes of biochemical metabolic markers in healthy young males - the Bispebjerg study of diurnal variations. Scand J Clin Lab Invest. 2015;75(8):686-92. doi: 10.3109/00365513.2015.1080385. Epub 2015 Sep 17. PMID 26378655
- [Background] Heegaard NH, Carlsen AL, Lilje B, Ng KL, Ronne ME, Jorgensen HL, Sennels H, Fahrenkrug J. Diurnal Variations of Human Circulating Cell-Free Micro-RNA. PLoS One. 2016 Aug 5;11(8):e0160577. doi: 10.1371/journal.pone.0160577. eCollection 2016. PMID 27494182
- [Background] Schroor MM, Sennels HP, Fahrenkrug J, Jorgensen HL, Plat J, Mensink RP. Diurnal Variation of Markers for Cholesterol Synthesis, Cholesterol Absorption, and Bile Acid Synthesis: A Systematic Review and the Bispebjerg Study of Diurnal Variations. Nutrients. 2019 Jun 26;11(7):1439. doi: 10.3390/nu11071439. PMID 31247945
- [Background] Rehfeld JF, Sennels HP, Jorgensen HL, Fahrenkrug J. Circadian variations in plasma concentrations of cholecystokinin and gastrin in man. Scand J Clin Lab Invest. 2020 Nov;80(7):546-551. doi: 10.1080/00365513.2020.1804072. Epub 2020 Aug 21. PMID 32820681
- [Derived] Zilstorff DB, Richter MM, Hannibal J, Jorgensen HL, Sennels HP, Wewer Albrechtsen NJ. Secretion of glucagon, GLP-1 and GIP may be affected by circadian rhythm in healthy males. BMC Endocr Disord. 2024 Mar 14;24(1):38. doi: 10.1186/s12902-024-01566-9. PMID 38481208